CLINICAL TRIAL: NCT02461472
Title: The Risk Analysis for Diabetic Cardiovascular Autonomic Neuropathy in General Chinese Population
Brief Title: Risk Analysis for Diabetic Cardiovascular Autonomic Neuropathy
Status: Completed | Type: Observational
Sponsor: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Collaborators: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Zihui Tang, M.D and Ph.D, Huashan Hospital
Other Study IDs: DCANRA_Dr.Tang
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Diabetic Cardiovascular Autonomic Neuropathy
Keywords: risk factors; risk analysis; diabetic cardiovascular autonomic neuropathy; general Chinese population

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Dr.Tang's research group: Dr.Tang's research group for clinical risk analysis of human complex disease
  Interventions: Other: not intervention

INTERVENTIONS:
Other: not intervention — This is a cross-sectional study, no intervention was performed.
  Other Names: nothing

SUMMARY:
A large-scale, community-based, cross-sectional study was conducted to explore the extent to which risk factors associated with diabetic cardiovascular autonomic neuropathy (DCAN) in general Chinese population. A total of more than 2000 diabetic participants were recruited by using multiple stages sampling (first cluster sampling and then simply sampling). Data involved in demographic information, clinical biomarkers such as glucose and lipids profiles, medical and therapy history were collected. Every participants was complete DNA extracted and genotyped. Diabetic Cardiovascular autonomic functions were measured by using short-term heart rate variability (HRV) to evaluate the outcome of DCAN. Univariate and multiple variables analysis have been performed to examine potential environmental and genetic risk factors of CAN. In addition, clinical risk model, simply screening model and nonlinear system model such as artificial neural network was created, respectively.

DETAILED DESCRIPTION:
Little is known about the risk factors and risk models for diabetic cardiovascular autonomic neuropathy in Chinese population. A large-scale, community-based, cross-sectional study was conducted to explore the extent to which risk factors associated with diabetic cardiovascular autonomic neuropathy (DCAN) in general Chinese population. A total of more than 2000 diabetic participants were recruited by using multiple stages sampling (first cluster sampling and then simply sampling). Data involved in demographic information, clinical biomarkers such as glucose and lipids profiles, medical and therapy history were collected. Every participants was complete DNA extracted and genotyped. Diabetic Cardiovascular autonomic functions were measured by using short-term heart rate variability (HRV) to evaluate the outcome of DCAN. Univariate and multiple variables analysis have been performed to examine potential environmental and genetic risk factors of CAN. In addition, clinical risk model, simply screening model and nonlinear system model such as artificial neural network was created, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Survey Chinese participants with undiagnosed DCAN Aged 30-90 years, were included in this study.

Exclusion Criteria:

* Some diabetic patients were excluded from the study to eliminate potential confounding factors that may have influenced their CA function. Briefly, the exclusion criteria were as follows:

  1. history or findings of arrhythmia and hyperthyroidism or hypothyroidism
  2. pregnancy or lactation
  3. serious hepatic or renal dysfunctions (GFR < 30 mL/min/1.73m2).

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators recruited participants from rural and urban communities in Shanghai. Survey diabetic participants with undiagnosed DCAN, aged 30-90 years, were included in this study. Our study invited a total of 3000 subjects to a screening visit between 2013 and 2015.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2013-01 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Autonomic Neuropathy (CAN) measured by short-term short-term heart rate variability (HRV) | participants will be measured for the duration of outpatient stay, an expected average of 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zihui Tang, M.D and Ph.D, Principal Investigator — Huashan Hospital
Locations (1):
- Huasha Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Li Z, Tang ZH, Zeng F, Zhou L. Associations between the severity of metabolic syndrome and cardiovascular autonomic function in a Chinese population. J Endocrinol Invest. 2013 Dec;36(11):993-9. doi: 10.3275/9005. Epub 2013 Jun 17. PMID 23770583
- [Result] Tang ZH, Zeng F, Li Z, Zhou L. A risk score of cardiovascular autonomic dysfunction for targeted screening in the Chinese population. Int J Cardiol. 2013 Oct 12;168(5):4861-2. doi: 10.1016/j.ijcard.2013.07.062. Epub 2013 Jul 25. No abstract available. PMID 23890865
- [Result] Tang ZH, Liu J, Zeng F, Li Z, Yu X, Zhou L. Comparison of prediction model for cardiovascular autonomic dysfunction using artificial neural network and logistic regression analysis. PLoS One. 2013 Aug 5;8(8):e70571. doi: 10.1371/journal.pone.0070571. Print 2013. PMID 23940593
- [Result] Tang ZH, Zeng F, Yu X, Zhou L. Bayesian estimation of cardiovascular autonomic neuropathy diagnostic test based on baroreflex sensitivity in the absence of a gold standard. Int J Cardiol. 2014 Feb 15;171(3):e78-80. doi: 10.1016/j.ijcard.2013.11.100. Epub 2013 Dec 6. No abstract available. PMID 24360155
- [Result] Tang ZH, Fang Z, Zhou L. Human genetics of diabetic vascular complications. J Genet. 2013 Dec;92(3):677-94. doi: 10.1007/s12041-013-0288-1. PMID 24371189
- [Result] Zeng F, Tang ZH, Li Z, Yu X, Zhou L. Normative reference of short-term heart rate variability and estimation of cardiovascular autonomic neuropathy prevalence in Chinese people. J Endocrinol Invest. 2014 Apr;37(4):385-91. doi: 10.1007/s40618-013-0047-4. Epub 2014 Jan 9. PMID 24633734
- [Result] Tang ZH, Zeng F, Li Z, Zhou L. Association and predictive value analysis for resting heart rate and diabetes mellitus on cardiovascular autonomic neuropathy in general population. J Diabetes Res. 2014;2014:215473. doi: 10.1155/2014/215473. Epub 2014 Mar 18. PMID 24772443
- [Result] Tang ZH, Wang L, Zeng F, Li Z, Yu X, Zhang K, Zhou L. Bayesian estimation of cardiovascular autonomic neuropathy diagnostic test based on short-term heart rate variability without a gold standard. BMJ Open. 2014 Oct 6;4(9):e005096. doi: 10.1136/bmjopen-2014-005096. PMID 25287103
- [Result] Zhang L, Tang ZH, Zeng F, Li Z, Zhou L, Li Y. Clinical risk model assessment for cardiovascular autonomic dysfunction in the general Chinese population. J Endocrinol Invest. 2015 Jun;38(6):615-22. doi: 10.1007/s40618-014-0229-8. Epub 2015 Jan 3. PMID 25555369
- [Derived] Song L, Zhou L, Tang Z. An association analysis of lipid profile and diabetic cardiovascular autonomic neuropathy in a Chinese sample. Lipids Health Dis. 2016 Jul 26;15:122. doi: 10.1186/s12944-016-0287-3. PMID 27457375
- [Derived] Ge X, Chen H, Zhang K, Tang ZH. The analysis of blood pressure profiles and their severity in relation to diabetic cardiovascular autonomic neuropathy in the Chinese population: preliminary analysis. J Endocrinol Invest. 2016 Aug;39(8):891-8. doi: 10.1007/s40618-016-0444-6. Epub 2016 Mar 3. PMID 26940214